CLINICAL TRIAL: NCT06878898
Title: Impact of a Mobile Phone and Educational Intervention on Health-related Quality of Life and Health Behaviors of African Americans With Asthma or COPD
Brief Title: Impact of a Mobile Phone and Educational Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kent State University (Other)
Responsible Party: Principal Investigator, Melissa Zullo, Professor and Interim Associate Dean, Kent State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 16-061
Record Dates: First submitted 2023-06-01; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Asthma COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Asthma COPD Workshop) and mobile phone (Experimental): The ACOPD Workshop comprised of 1-hour educational sessions on basic disease knowledge (one session) and management practices (two sessions). Participants were given:
  * devices and items to encourage behavioral change related to the intervention i.e., pedometers, pocket calendars (tracking physical activity) and pill boxes (medication adherence)
  * handouts on asthma, COPD developed based on the ACOPD Workshop content asthma and COPD action plan templates from the American Lung Association (ALA) and Asthma and Allergy Foundation of America (AAAF) to encourage dialogue with their healthcare provider, and
  * a certificate of completion for those that attended all three sessions.
    * The mobile text messaging provided informational support to reinforce the importance of the core health behaviors presented in the educational sessions. Participants in the intervention arm received text messages once per day over four weeks.
  Interventions: Behavioral: Education and mobile phone text-messaging
- Education only (Active Comparator): The ACOPD Workshop comprised of 1-hour educational sessions on basic disease knowledge (one session) and management practices (two sessions) i.e., three core health behaviors (nutrition, physical activity, and avoiding triggers) recommended for proper management of asthma and COPD. Participants were given:
  * devices and items to encourage behavioral change related to the intervention i.e., pedometers, pocket calendars (tracking physical activity) and pill boxes (medication adherence)
  * handouts on asthma, COPD developed based on the ACOPD Workshop content
  * asthma and COPD action plan templates from the American Lung Association (ALA) and Asthma and Allergy Foundation of America (AAAF) to encourage dialogue with their healthcare provider, and
  * a certificate of completion for those that attended all three sessions.
  Interventions: Other: Education only

INTERVENTIONS:
Behavioral: Education and mobile phone text-messaging — The investigators piloted a knowledge and mobile text-messaging intervention using a prospective group design, allocating 14 (asthma=8; COPD=6) and 15 (asthma=9; COPD=6) participants to control and intervention groups respectively, after stratifying by type of disease.
  Arms: Education (Asthma COPD Workshop) and mobile phone
Other: Education only — Participants in the control group only received the educational intervention.
  Arms: Education only

SUMMARY:
The purpose of this pilot study was to:

1. partner with African American churches to increase awareness of COPD.
2. use a community-based approach to facilitate early detection of COPD in the church setting. The pre-screening with a paper-based tool and spirometry testing were provided at community health fairs at the churches.
3. determine the impact of a combined intervention (education and mobile phone/text messages) on health related-related quality of life and health behaviors of African Americans with asthma and COPD.

The study used a randomized controlled trial (RCT) design to assess the effect of the intervention (education and mobile text-messaging) on health-related quality of life and health behaviors recommended for improved COPD self-management. All participants received the educational component then were randomized to a control group and intervention group, in which participants received mobile phone-based text messages on improving health behaviors associated with better self-management of asthma and COPD.

DETAILED DESCRIPTION:
This pilot study evaluated the feasibility and impact of a combined intervention on HRQOL and three health behaviors (nutrition, physical activity, avoiding triggers) in African Americans with asthma or COPD. This was a community-based intervention that recruited participants from six predominantly African American churches. African Americans over 18 years with asthma or COPD were randomized to control or intervention. Intervention received education (asthma COPD (ACOPD) Program) and a one-month text-messaging program, while control received the ACOPD Program alone. Measures were made at three- and 9-month follow-up. Independent and paired t-tests were used to examine HRQOL between groups and over time.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants for the study were African American adults of 18 years and above.

Participants had to have reported physician diagnosed (on the survey distributed at the church) or spirometry diagnosed (at the community health fair) asthma or COPD, access to a text-messaging enabled mobile phone, and provision of signed informed consent.

Exclusion Criteria:

* Individuals unwilling to participate in the study and patients with other chronic lung diseases, terminal, or comorbid illnesses more severe in nature than asthma or COPD (i.e., heart disease and cancer) were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Disease Knowledge: Knowledge and Management Questionnaire | Baseline, 3 months after ACOPD workshop, 9-months post-ACOPD workshop
  Disease Knowledge: A knowledge questionnaire on basic disease concepts and management practices
Health-related quality of life (HRQOL) in participants with Chronic Obstructive Pulmonary Disease (COPD) | Baseline, 3 months after ACOPD workshop, 9-months post-ACOPD workshop
  Health-related quality of life: The validated Clinical COPD Questionnaire used to measure HRQOL. The scores range from 0 to 6, higher values indicate poorer health status, and a change in score >0.4 is considered clinically important.
Health-related quality of life in participants with Asthma | Baseline, 3 months after ACOPD workshop, 9-months post-ACOPD workshop
  Health-related quality of life at baseline: The validated 15-item mini-Asthma Quality of Life Questionnaire (mAQLQ) used to measure HRQOL. The scores range from 1-7, higher scores indicate better health status, and a change in score >0.5 is considered clinically important.

SECONDARY OUTCOMES:
Respiratory management behaviors | Baseline, 3 months after ACOPD workshop, 9-months post-ACOPD workshop
  Respiratory Management Behaviors Questionnaire (RMBQ) at baseline: A study-developed questionnaire with 27 items and were summarized as frequencies and proportions.
Self-efficacy | Baseline, 3 months after ACOPD workshop, 9-months post-ACOPD workshop
  Self-Efficacy Questionnaire (SEQ) at baseline: The Self-Efficacy Questionnaire with 6-items from a combination of self-efficacy scales developed for chronic illness. The scale ranges from 1-10 and higher scores indicate higher self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Kent State University, Kent, Ohio, United States

IPD SHARING:
Plan to Share IPD: No